CLINICAL TRIAL: NCT00704327
Title: Evaluating the Impact of Cerebral Ischemic And Degenerative Changes On Cognition
Status: Terminated | Type: Observational
Why Stopped: Investigator left the Institution
Sponsor: Lahey Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 2008-029
Record Dates: First submitted 2008-06-20; First posted 2008-06-24 (Estimated); Last update posted 2017-12-21 (Actual); Status verified 2017-08

CONDITIONS: Cognitive Decline
Keywords: Cognitive Functions; Brain Ischemia; Cerebral Atrophy; Dementia; Intracranial atherosclerosis; Memory impairment
MeSH Terms: conditions — Cognitive Dysfunction; Brain Ischemia; Dementia; Intracranial Arteriosclerosis; Memory Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate whether or not cerebral atrophy scores obtained from a brain MRI can correlate with Cognitive Test results. These results hope to demonstrate a link between cerebral ischemic/degenerative changes shown on the MRI and cognition functions results.

DETAILED DESCRIPTION:
Preliminary evidence indicates that intracranial atherosclerosis may predict incident cerebrovascular events and central atrophy. Age induced changes on cerebral tissue in adulthood is witnessed as atrophy and well know ischemic changes on imaging studies. There is no consensus at this time what constitutes normal, age induced atrophy and pathologic atrophy on imaging studies. The same challenge is also encountered for ischemic cerebral parenchymal change.

Until recently there have been several important limitations in this research 1) Measurement of cerebral tissue loss and amount of ischemic insult was based on a qualitative grading (2) There was no cognitive testing. With Advancements in software technology that have now allowed for measurements of CSF and brain volumes in reliable and reproducible ways and the neuroradiologist having access to the subject's Neurological Cognitive Testing Scores, this study will objectively measure MRI findings and correlate them with the level of cognitive function.

This study will look at subjects who have undergone cognitive testing from the Neurology Clinic and then referred for an MRI brain exam, as standard of care testing. The MRI information will be acquired by volumetric technique for calculation of brain and CSF volumes and MRI data will be plotted against the cognitive test results.

The results of this study will be to correlate quantitative measures of cerebral atrophic and ischemic changes with level of cognition and to establish reliable imaging criteria that can help identify normal, age induced versus pathologic. Information obtained will shed light to cognitive effects and imaging appearance of: Separation of normal age related changes from pathologic states, changes leading to dementia and normal pressure hydrocephalus.

ELIGIBILITY:
Inclusion Criteria:

* Subjects older than 50 years of age
* Subjects who have undergone Cognitive Testing
* Subjects who can cooperate and give informed consent

Exclusion Criteria:

* Subjects with known medical conditions predisposing them for atrophy such as: Chronic renal failure, HIV, head/neck tumors, prior radiation, post- traumatic brain disorder, metabolic disorders of brain, polysubstance abuse, and steroid use

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects identified from Neurology Department who have already undergone Cognitive Testing and have been referred for an MRI exam
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2008-02 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Correlate quantitative measures of cerebral atrophic and ischemic changes with level of cognition using Mental Status Exam and Brain MRI exam | One time visit, duration of MRI

SECONDARY OUTCOMES:
Establish reliable imaging criteria to identify normal age induced changes versus pathologic process comparing Mental Status Exam with Brain MRI(measuring CSF and Brain volumes) | Duration of study 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Sami H. Erbay, M.D., Principal Investigator — Lahey Clinic, Inc.
Locations (1):
- Lahey Clinic, Inc., Burlington, Massachusetts, United States

REFERENCES:
- [Background] Ylikoski A, Erkinjuntti T, Raininko R, Sarna S, Sulkava R, Tilvis R. White matter hyperintensities on MRI in the neurologically nondiseased elderly. Analysis of cohorts of consecutive subjects aged 55 to 85 years living at home. Stroke. 1995 Jul;26(7):1171-7. doi: 10.1161/01.str.26.7.1171. PMID 7604409
- [Background] Kamata T, Hishida A, Takita T, Sawada K, Ikegaya N, Maruyama Y, Miyajima H, Kaneko E. Morphologic abnormalities in the brain of chronically hemodialyzed patients without cerebrovascular disease. Am J Nephrol. 2000 Jan-Feb;20(1):27-31. doi: 10.1159/000013551. PMID 10644864
- [Background] Muuronen A, Bergman H, Hindmarsh T, Telakivi T. Influence of improved drinking habits on brain atrophy and cognitive performance in alcoholic patients: a 5-year follow-up study. Alcohol Clin Exp Res. 1989 Feb;13(1):137-41. doi: 10.1111/j.1530-0277.1989.tb00298.x. PMID 2646967
- [Background] National Heart, Lung, and Blood Institute(NHLBI), National Institutes of Health. Morbidity and mortality: 2000 chart book on cardiovascular, lung and blood disease. Abailable at: http://www.nhlbi.nih.gov/resources/docs/00chtbk.pdf. Accessed February 13, 2002
- [Background] Knopman DS, Mosley TH, Catellier DJ, Sharrett AR; Atherosclerosis Risk in Communities (ARIC) Study. Cardiovascular risk factors and cerebral atrophy in a middle-aged cohort. Neurology. 2005 Sep 27;65(6):876-81. doi: 10.1212/01.wnl.0000176074.09733.a8. PMID 16186527
- [Background] Rumberger JA, Simons DB, Fitzpatrick LA, Sheedy PF, Schwartz RS. Coronary artery calcium area by electron-beam computed tomography and coronary atherosclerotic plaque area. A histopathologic correlative study. Circulation. 1995 Oct 15;92(8):2157-62. doi: 10.1161/01.cir.92.8.2157. PMID 7554196
- [Background] Arad Y, Spadaro LA, Goodman K, Lledo-Perez A, Sherman S, Lerner G, Guerci AD. Predictive value of electron beam computed tomography of the coronary arteries. 19-month follow-up of 1173 asymptomatic subjects. Circulation. 1996 Jun 1;93(11):1951-3. doi: 10.1161/01.cir.93.11.1951. PMID 8640967
- [Background] Arad Y, Spadaro LA, Goodman K, Newstein D, Guerci AD. Prediction of coronary events with electron beam computed tomography. J Am Coll Cardiol. 2000 Oct;36(4):1253-60. doi: 10.1016/s0735-1097(00)00872-x. PMID 11028480
- [Background] Wong ND, Hsu JC, Detrano RC, Diamond G, Eisenberg H, Gardin JM. Coronary artery calcium evaluation by electron beam computed tomography and its relation to new cardiovascular events. Am J Cardiol. 2000 Sep 1;86(5):495-8. doi: 10.1016/s0002-9149(00)01000-6. PMID 11009264
- [Background] Raggi P, Callister TQ, Cooil B, He ZX, Lippolis NJ, Russo DJ, Zelinger A, Mahmarian JJ. Identification of patients at increased risk of first unheralded acute myocardial infarction by electron-beam computed tomography. Circulation. 2000 Feb 29;101(8):850-5. doi: 10.1161/01.cir.101.8.850. PMID 10694523
- [Background] Simon A, Giral P, Levenson J. Extracoronary atherosclerotic plaque at multiple sites and total coronary calcification deposit in asymptomatic men. Association with coronary risk profile. Circulation. 1995 Sep 15;92(6):1414-21. doi: 10.1161/01.cir.92.6.1414. PMID 7664421
- [Background] Erbay S, Han R, Baccei S, Krakov W, Zou KH, Bhadelia R, Polak J. Intracranial carotid artery calcification on head CT and its association with ischemic changes on brain MRI in patients presenting with stroke-like symptoms: retrospective analysis. Neuroradiology. 2007 Jan;49(1):27-33. doi: 10.1007/s00234-006-0159-z. Epub 2006 Nov 7. PMID 17089112
- [Background] Babiarz LS, Yousem DM, Bilker W, Wasserman BA. Middle cerebral artery infarction: relationship of cavernous carotid artery calcification. AJNR Am J Neuroradiol. 2005 Jun-Jul;26(6):1505-11. PMID 15956522
- [Background] Yue NC, Arnold AM, Longstreth WT Jr, Elster AD, Jungreis CA, O'Leary DH, Poirier VC, Bryan RN. Sulcal, ventricular, and white matter changes at MR imaging in the aging brain: data from the cardiovascular health study. Radiology. 1997 Jan;202(1):33-9. doi: 10.1148/radiology.202.1.8988189.